CLINICAL TRIAL: NCT05447585
Title: A Prospective, Multicenter Clinical Trial of Coronary Atherectomy System in Patients With Calcified Coronary Artery Lesion
Brief Title: Coronary Atherectomy System in Patients With Coronary Calcification (CORECT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai MicroPort Rhythm MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMD-D-001
Record Dates: First submitted 2022-06-16; First posted 2022-07-07 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Calcification of Coronary Artery
Keywords: calcification, coronary artery
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronary Atherectomy System (Experimental): Subjects in experimental arm will be treated with the Coronary Atherectomy System manufactured by Shanghai Microport Rhythm Co. Ltd.
  Interventions: Device: Coronary atherectomy system of Shanghai MicroPort Rhythm
- Rotablator Rotational Atherectomy System (Active Comparator): Subjects in control arm will be treated with Rotablator Rotational Atherectomy System manufactured by Boston Scientific Corporation
  Interventions: Device: Rotablator Rotational Atherectomy System

INTERVENTIONS:
Device: Coronary atherectomy system of Shanghai MicroPort Rhythm — Coronary Atherectomy System utilizes a diamond-coated eccentric crown to expand the lumen diameter via centrifugal forces while rotating over an atherectomy guide wire.
  Other Names: Stenting will be applied in both arms
  Arms: Coronary Atherectomy System
Device: Rotablator Rotational Atherectomy System — The Rotablator Rotational Atherectomy System is comprised of a Rotablator RotaGlide, a Rotablator RotaLink Plus/RotaWire/Console
  Other Names: Stenting will be applied in both arms
  Arms: Rotablator Rotational Atherectomy System

SUMMARY:
This is a prospective and multicenter clinical investigation aiming to evaluate the safety and effectiveness of coronary atherectomy system for the treatment of patients with coronary calcification.

DETAILED DESCRIPTION:
This study is divided into two phases. The first phase is the pilot study stage, which is a prospective single group observational test (FIM stage). The second phase is the pivotal study phase, which is a prospective, multicenter, randomized controlled and non inferiority test (RCT phase). It is carried out in about 25 hospitals in China.

1. Pilot study phase (FIM phase): It is a prospective, multicenter and single-arm observational test. It is expected to recruit 15 subjects in 3 to 5 research centers in China. The primary endpoint is procedural success rate.
2. Pivotal study phase (RCT phase): It is a prospective, multicenter, randomized controlled and non inferiority trial. 224 subjects are expected to be recruited in 25 research centers in China and randomly divided into two groups according to the ratio of test group: control group = 1:1. The primary endpoint of the RCT phase is the rate of no major adverse cardiovascular events (MACE) at 30 days after baseline.
3. All subjects with coronary calcified lesions participating in this clinical study must have a calcified lesion length of no more than 40 mm and located in an coronary artery with a diameter of ≥ 2.50 mm but ≤ 4.00 mm.
4. All subjects receive clinical follow-up during hospitalization and 30 days, 6 months and 12 months after surgery.
5. Successful enrollment: The atherectomy guidewires pass through the target lesion successfully (through the true lumen), and there are no vascular perforation, dissection, thrombosis and other complications.

ELIGIBILITY:
Clinical Inclusion Criteria:

CI1. Age between 18 and 80.

CI2. Subjects who are going to accept percutaneous coronary intervention (PCI) and drug-eluting stent implantation.

CI3. Asymptomatic evidence of ischemia, stable or unstable angina pectoris, or old myocardial infarction.

CI4. Acceptable candidates for coronary artery bypass grafting (CABG).

CI5. The left ventricular ejection fraction (LVEF) is equal to or greater than 30% measured by echocardiography or left ventricle contrast examination within 30 days before inclusion.

CI6. Subjects who are able to understand the purpose of the trial, participate voluntarily or by proxy and indicate by signing the informed consent form that they recognize the risks and benefits described in the informed consent document and are willing to undergo clinical follow-up.

Angiography Inclusion Criteria:

AI1. There is only one target lesion that needs to be treated.

AI2. The target vessel must be a native coronary artery with reference diameter >= 2.5mm and <= 4.0 mm.

AI3. The target vessel must be with a stenosis of >= 70% and < 100%Target lesion angiographic stenosis, or of >=50% and <70% with local ischemic symptoms.

AI4. Target lesion length ≤ 40 mm .

AI5. The target lesion must have evidence of severe calcium deposit, or moderate calcification which cannot be fully expanded by PTCA balloon catheter at the lesion site based on the protocol criterion, .

Clinical Exclusion Criteria:

CE1. Acute myocardial infarction within 30 days prior to baseline procedure.

CE2. NYHA or Killip class III or IV heart failure.

CE3. Severe cardiac insufficiency with reduced ejection fraction (left ventricular ejection fraction < 30%).

CE4. Intracardiac thrombus within 30 days before inclusion.

CE5. Subjects who have received organ transplantation or is waiting for organ transplantation.

CE6. Subjects who are receiving chemotherapy or scheduled to receive chemotherapy 30 days before or after baseline surgery.

CE7. Subjects who are receiving chronic (≥ 72 hours) anticoagulant therapy (e.g. heparin, warfarin, coumarin) for indications other than acute coronary syndrome.

CE8. Participants' platelet < 50 × 10^9 / L or > 700 × 10^9 / L, and / or hemoglobin < 70g / L.

CE9. Subjects with confirmed or suspected liver diseases, including active hepatitis, or abnormal laboratory results are not suitable for the study.

CE10. Subjects diagnosed with chronic renal failure or has a serum creatinine level >2.5 mg/dl (or 221 µmol / L).

CE11. Subjects who have clear bleeding tendency, contraindications of antiplatelet preparation and anticoagulant treatment, and are unable to receive antithrombotic treatment.

CE12. History of cerebrovascular accident (CVA), transient ischemic attack (TIA), active peptic ulcer disease, gastrointestinal (GI) bleeding, transient ischemic attack (TIA), or permanent neurological defects that may lead to non-compliance with the test protocol in the past 6 months.

CE13. Target vessels (including collateral vessels) received any stent implantation within 12 months before baseline surgery.

CE14. Non target vessels were treated with any type of PCI within 24 hours before baseline surgery.

CE15. PCI or CABG is planned within 2 months after baseline procedure.

CE16. History of coronary endovascular brachytherapy at any time.

CE17. Known hypersensitivity to any drugs required by the stent or protocol (such as rapamycin or structure related compounds, fluoropolymers, aspirin or tigrelol, contrast medium, acrylic acid, stainless steel, chromium, nickel, iron, tungsten).

CE18. Subjects who have other serious medical diseases (such as cancer, congestive heart failure), which may reduce life expectancy to less than 12 months or it is expected to be difficult to complete 12-months follow-up.

CE19. Subjects who currently abuse drugs, such as heroin, alcohol, etc.

CE20. Subjects who plan to undergo surgery that may lead to non-compliance with the protocol or confusion in data interpretation.

CE21. Currently enrolled in any other clinical trial (does not reach its primary endpoint), or intended to participate in any other clinical trial within 12 months after baseline procedure.

CE22. Females subjects who are pregnant,breast feeding or planning to become pregnant within the study period.

CE23. Untrolled diabetes.

CE24. Inability to understand the study or a history of non-compliance with medical advice.

Angiographic Exclusion Criteria:

AE1. Target lesions that meet the following criteria:

* Ostial lesions (within 5mm of ostium);
* Target lesions involve bifurcation lesions, and branch vessels need to be implanted with stents;
* Angular lesions (> 45 °)
* Located in a native vessel distal to anastomosis with a saphenous vein graft or LIMA/RIMA bypass;
* Thrombosis in the target vessel;
* Target lesion dissection;
* In-stent restenosis;
* Chronic total occlusion lesions that cannot be passed through by atherectomy guidewire.

AE2. Unprotected left main coronary artery disease (> 50% diameter stenosis).

AE3. Protected left main coronary artery disease (> 50% diameter stenosis at LMCA and left coronary artery receive bypass grafting), and the target lesion is located in LAD or LCX.

AE4. Other clinical significant lesions in target vessels may require intervention within 2 months after baseline surgery.

AE5. The target vessel (including collateral) near the target lesion or within 10 mm (visually) from the distal end of the target lesion has received stent implantation at any time before baseline surgery.

AE6. Especially tortuous target vessels. AE7. Non-target lesion failed to be treated before the treatment of target lesion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
FIM phase: Clinical success | During hospitalization (up to 7 days after baseline procedure).
  Clinical success is defined as successful stent delivery with a residual stenosis of <50% and TIMI flow III without adverse events during procedure the occurrence of an in-hospital MACE (up to 7 days after surgery).
RCT phase: 30-Day Freedom From Major Adverse Cardiac Events (MACE) | 30 days after baseline procedure.
  MACE is composed of cardiac death, myocardial infarction and target vessel revascularization.

SECONDARY OUTCOMES:
Device success | Baseline procedure
  Device success is defined as successful stent delivery after atherectomy and without periprocedural complications
Procedural success | Baseline procedure
  Procedural success was defined as successful stent delivery with <50% residual stenosis and TIMI flow III and without periprocedural complications
Procedure-related complications | Baseline procedure
  Procedure-related complications are defined as severe dissection (Type D to F), perforation, stent upload and in-stent thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, M.D., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China